CLINICAL TRIAL: NCT01169883
Title: Coping Peer Intervention for Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Giselle Mosnaim, Principal Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 09111001; 1R21HL098812-01A1 (NIH)
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: adherence; asthma; pediatrics; behavioral intervention; inner city
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Control Group (Active Comparator): 1) Doctor Asthma Messages delivered over a 10 week time period; 2) Asthma Supervision; and 3) Music Tracks.
  Interventions: Behavioral: Doctor Asthma Messages; Behavioral: Asthma Supervision; Behavioral: Music Tracks
- Intervention Group (Experimental): 1) Coping Peer Support delivered over a 10 week time period; 2) Coping Peer Asthma Messages delivered over a 10 week time period; 3) Asthma Supervision; and 4) Music Tracks.
  Interventions: Behavioral: Coping Peer Support; Behavioral: Coping Peer Asthma Messages; Behavioral: Asthma Supervision; Behavioral: Music Tracks

INTERVENTIONS:
Behavioral: Coping Peer Support — The Coping Peer Support is delivered at weekly group meetings over the 10 week active treatment phase. The Coping Peer Support consists of: group support, coping peer group problem solving, and development and recording of Coping Peer Asthma Messages. More specifically, a social worker facilitates a peer group discussion of barriers to taking their daily inhaled steroids, and ways to overcome these barriers. The social worker also facilitates peer recording of messages by the participants encouraging each other to take their daily inhaled steroid medication.
  Arms: Intervention Group
Behavioral: Doctor Asthma Messages — The attention control group will receive Doctor Asthma Messages delivered during the 10 week active treatment phase. The content and number of these messages will be equivalent to those received by the intervention group. These messages are developed and recorded by an Allergist/Immunologist. The participants in the attention control group will listen to these Doctor Asthma Messages, between their favorite music tracks on their MP3 player, as they go about their day-to-day activities.
  Arms: Attention Control Group
Behavioral: Coping Peer Asthma Messages — The Coping Peer Asthma Messages developed and recorded by study participants for each other at the weekly coping peer group meetings will be placed on intervention group participants' MP3 players. These Coping Peer Asthma Messages will be played on their MP3 players, between their favorite music tracks, during the course of their daily routines. This infuses the coping peer support from the coping peer group meetings into the adolescents' daily routines.
  Arms: Intervention Group
Behavioral: Asthma Supervision — A member of the study team meets individually with each participant at baseline to teach proper use of a peak flow meter and spacer.
Behavioral: Music Tracks — Participants receive an MP3 player (iPod Shuffle) in the baseline period. Participants receives clean, radio-edited music tracks of their choice in the baseline period and 10 week active treatment period.

SUMMARY:
Inner-city African American and Hispanic adolescents suffer from disproportionately high rates of emergency room visits and hospitalizations for acute exacerbations of asthma. This study proposes the use of a coping peer support intervention, enhanced by a technology-based platform that infuses peer support throughout adolescents' daily routines, to increase adherence to daily controller medications and ultimately reduce asthma exacerbation risk in this important population subgroup.

DETAILED DESCRIPTION:
High rates of asthma morbidity and mortality among inner-city African American and Hispanic adolescents demand urgent intervention. To address this disparity, the investigators have designed a culturally sensitive intervention aimed at improving adherence to daily controller medications for asthma, and ultimately reduce asthma exacerbation risk, that fits easily into adolescents' chaotic lifestyles.

The proposed study is a behavioral randomized controlled trial that tests if a coping peer intervention can increase adherence to asthma controller medications among urban African American and Hispanic adolescents 11 to 16 years of age. To ensure the project's success, the principal investigator has assembled a multi-disciplinary team of researchers, including behavioral and social science experts. The Specific Aims propose to: (1) evaluate the impact of a 10-week coping peer support intervention on adherence and knowledge, compared to an attention control; (2) evaluate the ability of a 10-week coping peer support intervention to achieve sustained post-treatment improvements in adherence and knowledge, compared to an attention control; and (3) to develop estimates needed for the design of a subsequent R01 behavioral controlled trial testing the efficacy of this intervention to decrease risk of asthma exacerbations. The study's primary outcome is adherence to daily asthma controller medications, measured using an objective electronic monitor. Study participants will be randomized to receive equal asthma supervision and music tracks plus either: (1) group support, coping peer group problem solving, and peer delivered asthma messages (intervention group); or (2) study team developed and recorded asthma health messages (attention control group) between music tracks, on a portable MP3 player. The group support and coping peer group problem solving consists of: putting subjects together in a small group to discuss barriers to adherence and ways to overcome these barriers; then having group members record messages to each other about overcoming barriers that will be played on their MP3 player, between music tracks, during the course of their daily routines. This effectively brings the coping peer support from the group into the course of the adolescents' day-to-day lives. The investigators hypothesize that it is the ability of the MP3 player to facilitate ongoing peer support that will be the basis for improved adherence. The long term goal is to apply the data from this research to submit an R01 grant application to conduct a behavioral randomized trial evaluating the effectiveness of this coping peer intervention to improve adherence, and ultimately reduce asthma exacerbations, in urban African American and Hispanic adolescents with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American or Hispanic
* 11-16 years of age
* Have persistent asthma
* Be on a prescription daily inhaled steroid medication for asthma

Exclusion Criteria:

* Candidate refusal
* Presence of other co-morbidities that could interfere with study participation
* greater than 47% adherence to daily inhaled steroid medication as measured at baseline using the Doser CT

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Objectively measured adherence to inhaled corticosteroids using an electronic dose counter, (Doser CT; Meditrac, Inc., Hudson, MA) | 10 weeks
  Adherence is measured as the average of daily adherence to prescribed inhaled corticosteroid medication dose over 14 days at both baseline and at 10 weeks. The average rate of adherence in the intervention group at 10-weeks will be compared to that in the attention control group, adjusting for baseline levels, using a hierarchical linear model since participants are clustered into groups.

SECONDARY OUTCOMES:
Asthma Knowledge assessed using the ZAP Asthma Knowledge Instrument | 10 weeks
  The average score on the ZAP Asthma Knowledge Instrument in the intervention group at 10-weeks will be compared to that in the attention control group, adjusting for baseline levels, using a hierarchical linear model since participants are clustered into groups.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle S Mosnaim, MD, MS, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States